CLINICAL TRIAL: NCT06311903
Title: Is Low Dose Norepinephrine Effective in Preperiod of Hypotensive Resuscitation in Hemorrhagic Shock?
Brief Title: Norepinephrine in Preperiod of Hypotensive Resuscitation in Hemorrhagic Shock
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rabab Mohamed Mohamed Mohamed, Assistant Professor of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36264PR430/11/23
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Norepinephrine; Hemorrhagic Shock; Hypotensive Resuscitation
MeSH Terms: conditions — Shock, Hemorrhagic | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Patients were received resuscitative fluid [administered at beginning with the arrival of the patient in the emergency department (mean blood pressure >70 mmHg)] followed by low dose of norepinephrine (NE) (0.05-0.2 μg/kg/min).
  Interventions: Drug: Low dose of Norepinephrine (NE)
- Group II (Experimental): patients were received resuscitative fluid. If there were no response to treatment to resuscitative fluid, they received norepinephrine (NE) gradually till reach high dose (≥0.3 μg/kg/min).
  Interventions: Drug: High dose of Norepinephrine (NE)

INTERVENTIONS:
Drug: Low dose of Norepinephrine (NE) — Patients were received resuscitative fluid [administered at beginning with the arrival of the patient in the emergency department (mean blood pressure >70 mmHg)] followed by low dose of NE (0.05-0.2 μg/kg/min).
  Arms: Group I
Drug: High dose of Norepinephrine (NE) — Patients were received resuscitative fluid. If there were no response to treatment to resuscitative fluid, they received NE gradually till reach high dose (≥0.3 μg/kg/min).
  Arms: Group II

SUMMARY:
The aim of this work was to investigate the effects of low dose of norepinephrine in preperiod of hypotensive resuscitation in hemorrhagic shock.

DETAILED DESCRIPTION:
Hemorrhagic shock is one of the leading causes of death following trauma. New fluid resuscitation concepts, including hypotensive, hypothermic, and delayed resuscitation for uncontrolled hemorrhagic shock, have been put forward and obtained a good effect both in clinical and laboratory parameters. The 2019 European guideline on the management of major bleeding and coagulopathy following trauma recommends the use of norepinephrine (NE) for maintaining target arterial blood pressure in patients with life-threatening hypotension. NE has potent α-adrenergic receptor activation activity, which can stimulate α-1 adrenergic receptors on peripheral vascular smooth muscles. High-dose NE may result in excessive arteriolar vasoconstriction which subsequently leads to the disorder of microcirculation and tissue hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Both sexes.
* Patients with hemorrhagic shock

Exclusion Criteria:

* Patients with cardiac arrest at admission.
* Severe brain.
* Spinal injury (because of different target blood pressures).
* Death due to hemostatic failure within 6 h of admission.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
24 hours mortality | 24 hours after intervention
  24 hours mortality will be measured.

SECONDARY OUTCOMES:
28 day mortality | 28 days after intervention
  28 day mortality will be measured.
Incidence of acute kidney injury | 24 hours after intervention
  Incidence of acute kidney injury will be measured within 24 hours.
Length of hospital stay | 28 days after intervention
  Length of hospital stay will be measured from admission till hospital discharge.
Length of intensive care unit stay | 28 days after intervention
  Length of intensive care unit (ICU) stay will be measured from admission till intensive care discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.